CLINICAL TRIAL: NCT05594134
Title: Efficacy of an Automatic Toothbrush With Nylon Bristles in Removing Dental Plaque: a Randomized Cross-over Study
Brief Title: Efficacy of an Automatic Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Lorenzo Franchi, Professor, University of Florence
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IUFET2
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Automatic toothbrush with nylon bristles (Experimental)
  Interventions: Other: Automatic toothbrush with nylon bristle
- Automatic toothbrush with silicone bristles (Active Comparator)
  Interventions: Other: Automatic toothbrush with silicone bristle
- Manual toothbrush used for 2 minutes (Active Comparator)
  Interventions: Other: Manual toothbrush used for 2 minutes
- Manual toothbrush used for 45 seconds (Active Comparator)
  Interventions: Other: Manual toothbrush used for 45 seconds
- No brushing (No Intervention)

INTERVENTIONS:
Other: Automatic toothbrush with nylon bristle — The automatic toothbrush with nylon bristles will be used for 10 seconds per dental arch
  Arms: Automatic toothbrush with nylon bristles
Other: Automatic toothbrush with silicone bristle — The automatic toothbrush with silicone bristles will be used for 10 seconds
  Arms: Automatic toothbrush with silicone bristles
Other: Manual toothbrush used for 2 minutes — A conventional manual toothbrush will be used for 2 minutes
  Arms: Manual toothbrush used for 2 minutes
Other: Manual toothbrush used for 45 seconds — A conventional manual toothbrush will be used for 45 seconds
  Arms: Manual toothbrush used for 45 seconds

SUMMARY:
The objective of this study is to compare the efficacy in terms of bacterial plaque removal, in a single use, of a new Y-shaped automatic electric toothbrush with nylon bristles, compared with the electric toothbrush of similar shape but with silicone bristles, with the manual toothbrush, and with a negative control (no brushing) in a group of volunteer students.

Primary endpoint: difference in "full mouth plaque score" between before and after brushing.

Secondary endpoint: sensation of "clean mouth" assessed on VAS scale from 0 to 10 where 0 indicates no sensation of clean mouth and 10 maximum sensation of clean mouth.

Single-center, randomized, controlled, superiority, cross-over, examiner-blinded study with 5 treatments (Y-shaped electric toothbrush with nylon bristles, similarly shaped electric toothbrush with silicone bristles, manual brushing for 45 seconds, manual brushing for 2 minutes, no brushing), carried out in a single session and spaced one week apart.

ELIGIBILITY:
Inclusion Criteria:

* Absence of fixed orthodontic appliances
* Presence of at least 20 teeth
* Full mouth plaque score greater than 40%
* Having provided signed and dated informed consent.

Exclusion Criteria:

* Subjects with manual inability to perform normal oral hygiene maneuvers
* Subjects allergic to silicone or nylon.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Change in full mouth plaque score | 5 minutes
  Difference in full mouth plaque score between before and after brushing

SECONDARY OUTCOMES:
Perception of "clean mouth" | 5 minutes
  Sensation of "clean mouth" assessed on a visual analogue scale from 0 to 10 where 0 indicates no sensation of clean mouth and 10 maximum sensation of clean mouth

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, The University of Florence, Florence, Italy

IPD SHARING:
Plan to Share IPD: No